CLINICAL TRIAL: NCT07336797
Title: Role of Empagliflozin in Metabolic Changes Associated With Antiretroviral Therapy in Human Immunodeficiency Virus
Brief Title: Effect of Empagliflozin on Metabolic Outcomes in Adults Living With HIV Receiving Dolutegravir-Based Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrahman Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Mahmoud, Teaching and Research Assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL(3828)
Record Dates: First submitted 2025-11-20; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome; Obesity & Overweight; HIV (Human Immunodeficiency Virus)
Keywords: Obesity; Empagliflozin; PLWH; HIV; SGLT-2 inhibitor; Metabolic Syndrome; Weight
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight; Acquired Immunodeficiency Syndrome; Body Weight | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: This is a Phase II, single-center, parallel-group, randomized, double-blind, controlled study design. PWH will be recruited from the Cairo University HIV Clinic.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients in the control group will receive an identical placebo and Standard Antiretroviral Therapy (ART)
  Interventions: Drug: Placebo
- EMPA Group + SOC (Experimental): Patients in the intervention arm will receive Empagliflozin 10 mg once daily for 6 months in addition to the standard DTG-based antiretroviral therapy.
  Interventions: Drug: Empagliflozin (oral)

INTERVENTIONS:
Drug: Empagliflozin (oral) — Empagliflozin is an oral medication used primarily to treat type 2 diabetes. It belongs to a class of drugs called SGLT2 inhibitors (sodium-glucose co-transporter 2 inhibitors). Empagliflozin blocks SGLT2 proteins in the kidneys.
  This prevents glucose reabsorption, causing excess sugar to be excreted in urine.
  It helps lower blood sugar levels and can also reduce body weight and blood pressure.
  Other Names: Mellitofix 10 mg
  Arms: EMPA Group + SOC
Drug: Placebo — TDF/FTC+DLG
  Other Names: Group A; Inactive Substance
  Arms: Control Group

SUMMARY:
We investigate the role of empagliflozin in the treatment of obesity in PLWH.

DETAILED DESCRIPTION:
HIV remains a major global public health concern. In 2024, approximately 40.8 million people were living with HIV worldwide. Around 630,000 deaths occurred due to AIDS-related illnesses. The preferred first-line ART regimen includes: Tenofovir disoproxil fumarate (TDF)+Emtricitabine (FTC) or Lamivudine (3TC)+Dolutegravir (DTG).

The introduction of highly active antiretroviral therapy transformed HIV from a fatal disease into a manageable chronic condition, significantly reducing morbidity and mortality.

Integrase strand transfer inhibitors (INSTIs), particularly dolutegravir (DTG), have been associated with greater weight gain compared with non-INSTI antiretroviral regimens.

The observed weight gain is strongly linked to adverse metabolic outcomes, including increased incidence of metabolic syndrome, higher rates of insulin resistance, and dyslipidemia.

Individuals living with HIV receiving antiretroviral therapy (ART) have been shown to have approximately 1.5-fold higher odds of developing metabolic syndrome (MetS).

Over the long term, these alterations contribute to a significantly elevated risk of cardiovascular disease, including myocardial infarction and stroke.

Evidence from biopsy-based studies further demonstrates a substantial burden of (NAFLD), (NASH), and liver fibrosis among people living with HIV (PLWH).

On the other hand, Sodium-glucose co-transporter-2 (SGLT2) inhibitors have demonstrated:

Cardiovascular benefits: Reduction in major adverse cardiovascular events in patients with atherosclerotic disease, including those with hypertension, dyslipidemia, and obesity.

Metabolic control: Improved glycemia via renal glucose reabsorption inhibition, lowering hyperglycemia with minimal hypoglycemic risk.

Weight and metabolic effects: Reduced body weight, BMI, SBP, visceral adiposity, insulin resistance, improved oral glucose tolerance test (OGTT) values and fasting insulin, even in non-diabetic individuals.

Hepatic outcomes: Significant reduction in liver fat content in metabolic disorders, mediated by improved lipid metabolism, insulin sensitivity, and reduced hepatic inflammation, supporting metabolic dysfunction-associated steatotic liver disease (MASLD) management.

These combined effects make SGLT2 inhibitors a promising therapeutic option for addressing the multiple facets of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years up to 65 years old.
* Body Mass Index (BMI) > 30 kg/m^2.
* Currently receiving an integrase strand transfer inhibitor (INSTI)-based regimen (dolutegravir-based ART).
* Sustained virologic suppression, defined as HIV-1 RNA < 200 copies/mL for at least 6 months.
* Current CD4 count > 250 cells/mL.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus, defined as a fasting blood glucose level > 126 mg/dL or glycated hemoglobin (HbA1c) > 6.5% (or per ADA definition).
* Renal impairment (e.g., eGFR < 60 ml/min/1.73m^2).
* Active viral hepatitis B or C.
* Hypersensitivity to empagliflozin or any of its excipients.
* Pregnancy or breastfeeding.
* Current use of other SGLT-2 inhibitors.
* Drugs that may interact with empagliflozin (e.g., rifampin or phenytoin) or dolutegravir (e.g., antacids, carbamazepine, or phenytoin).
* Current or recent use of medications known to be associated with significant weight gain (e.g., systemic corticosteroids, antipsychotics, mood stabilizers, or other agents with established weight-promoting effects).
* Known thyroid disease, defined as TSH > 6.0 mIU/L or < 0.35 mIU/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Weight change | 6 months
  Weight will be measured in kilograms using a calibrated scale from baseline to 6 months in PLWH on dolutegravir-based antiretroviral therapy.

SECONDARY OUTCOMES:
Change in Total Cholesterol | 6 months
  Effects of empagliflozin versus placebo on Concentration of total cholesterol in serum, measured in mg/dL.
Change in Fasting Blood Glucose | 6 months
  Concentration of glucose in blood plasma, measured in mg/dL after a minimum 8-hour overnight fast.
Change in Glycated Hemoglobin (HbA1c) | 6 months
  The percentage of glycated hemoglobin in the blood, used as an indicator of long-term glycemic control.
Change in Serum Creatinine | 6 months
  Concentration of creatinine in the blood, measured in mg/dL
Change in Systolic and Diastolic Blood Pressure | 6 months
  Measured in millimeters of mercury (mmHg) while the participant is in a seated position. at baseline, 3 and 6 months.
Change in Body Mass Index (BMI) | Baseline and 6 months
  BMI is a calculation of body weight relative to height. It will be calculated as weight in kilograms divided by the square of height in meters (kg/m^2).
Change in Waist Circumference | Baseline, 3 and 6 months
  Waist circumference will be measured using a non-stretchable flexible tape measure. The measurement will be taken at the midpoint between the lowest rib and the iliac crest (top of the hip bone) while the participant is standing and at the end of a normal expiration. Measurements will be recorded in centimeters.
Change in Absolute CD4+ T-cell Count | baseline and 6 months
  The absolute number of CD4+ T-lymphocytes will be measured in peripheral blood using flow cytometry. Results will be reported in cells per cubic millimeter (cells/mm³).
Change in Plasma HIV-1 RNA Viral Load | baseline and 6 months
  Viral load will be quantified using a Real-Time Polymerase Chain Reaction (RT-PCR) assay. Results will be reported in copies per milliliter (copies/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Abbassi, Prof., Study Director — Cairo University; Abedalrahman Dosoky, Principal Investigator — Cairo University; Ahmed Kamel, Study Director — Cairo University
Locations (1):
- Faculty of Pharmacy, Cairo University | Kasr El-Aini, Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 months